

1 2 3 Lidocaine and ketamine levels in plasma after simultaneous lidocaine/ketamine infusions. An observational assessment of therapy effects and side-effects. 4 5 6 7 8 Research legislation: Ordinance on human research with the exception of Clinical trials (HRO). 9 10 Type of Research Project: Research project involving human subjects 11 12 13 14 Risk Categorisation: Category A 15 16 17 Sponsor Investigator: Wilhelm Ruppen, Prof. Head of the Pain Unit 18 19 Department of Anaesthesiology 20 University Hospital of Basel (USB) 21 Spitalstrasse 21 22 CH - 4031 Basel 23 Phone: +41 61 328 64 96 24 Fax: +41 61 265 57 20 25 E-mail: wilhelm.ruppen@usb.ch 26 27 28 29 Project Leader and PI: Tobias Schneider, MD 30 Senior Physician 31 Department of Anaesthesiology University Hospital of Basel (USB) 32 33 Spitalstrasse 21 CH - 4031 Basel 34 35 Phone: +41 61 328 65 43 36 Fax: +41 61 265 57 20 37 E-mail: tobias.schneider@usb.ch 38

| 39<br>40 | PROTO | OCOL SIG | GNATURE FORM | | |
|---|---|---|---|---|---|
| 41<br>42 | Study | Title | Lidocaine and ketamine levels in plasma after simultaneous lidocaine/ketamine infusions. An observational assessment of therapy effects and side-effects. | | |
| 43<br>44<br>45<br>46<br>47 | hereby<br>version | The project leader has approved the protocol version <b>[1.1 (dated 02.05.2023)]</b> and confirms hereby to conduct the project according to the protocol, the Swiss legal requirements, current version of the World Medical Association Declaration of Helsinki and the principles and procedures for integrity in scientific research involving human beings. | | | |
| 48<br>49 | Sponso | Sponsor Investigator: | | | |
| 50 | Name: | Wilhelm | Ruppen, Prof. | | |
| 51<br>52 | Date: | 8th of M | lay 2023 | Signature: | |
| 53 | | | | | |
| 54<br>55 | Project | Leader a | nd Principal Investigator: | | |
| 56 | Name: | Tobias S | chneider, MD | | |
| 57<br>58 | Date: | 08.05. | 2023 | Signature: | |
| 59<br>60 | Co-Inve | estigators | : | | |
| 61<br>62 | Name: | Flavia Fl | epp, pract. med. | | |
| 63<br>64 | Date: | 08.05. | 2023 | Signature: | F. Flyg |
| 65<br>66 | Name: | Matthijs o | de Leeuw, pract. med. | | |
| 67<br>68 | Date: | 08.05. | 2023 | Signature: | M. de hur |
| 69<br>70 | Name: | Regula S | Steiner, Dr. sc. nat. | | |
| 71 | Date: | 5.5.202 | 23 | Signature: | Regula Steiner |
| | | | | | <b>→</b> |

# **TABLE OF CONTENTS**

73

| 74 | TA | ABLE OF CONTENTS | 3 |
|---|---|---|---|
| 75 | Gl | LOSSARY OF ABBREVATIONS | 4 |
| 76 | Sī | TUDY SYNOPSIS | 5 |
| 77 | 1 | BACKGROUND AND PROJECT RATIONALE | 11 |
| 78 | 2 | PROJECT OBJECTIVES AND DESIGN | 12 |
| 79 | | 2.1 Hypothesis and primary objective | 12 |
| 80 | | 2.1.2 Secondary objectives | 12 |
| 81 | | 2.2 Primary and secondary endpoints | 12 |
| 82 | | 2.3 Project design | 13 |
| 83 | 3 | PROJECT POPULATION AND STUDY PROCEDURES | 13 |
| 84 | | 3.1 Project population, inclusion and exclusion criteria | 13 |
| 85 | | 3.2 Recruitment, screening and informed consent procedure | 14 |
| 86 | | 3.3 Study procedures | 14 |
| 87 | | 3.3.1 Investigated variables | 15 |
| 88<br>89 | | 3.3.2 Standard Procedure of lidocaine-ketamine infusions at the Pain USB | Unit of<br>16 |
| 90 | | 3.3.3 Laboratory Analysis | 16 |
| 91 | | 3.4 Withdrawal and discontinuation | 16 |
| 92 | 4 | STATISTICS AND METHODOLOGY | 17 |
| 93 | | 4.1. Statistical analysis plan | 17 |
| 94 | | 4.2. Handling of missing data | 17 |
| 95 | 5 | REGULATORY ASPECTS AND SAFETY | 18 |
| 96 | | 5.1 Local regulations / Declaration of Helsinki | 18 |
| 97 | | 5.2 Notification of safety and protective measures (HRA Art. 15, HRO Art. 20) | 18 |
| 98 | | 5.3 Serious events (HRO Art. 21) | 18 |
| 99 | | 5.4 Amendments | 18 |
| 100 | | 5.5 End of project | 18 |
| 101 | | 5.6 Insurance | 18 |
| 102 | 6 | FURTHER ASPECTS | 18 |
| 103 | | 6.1 Overall ethical considerations | 18 |
| 104 | | 6.2 Risk-Benefit Assessment | 19 |
| 105 | 7 | QUALITY CONTROL AND DATA PROTECTION | 19 |
| 106 | | 7.1 Quality measures | 19 |
| 107 | | 7.2 Data recording and source data | 19 |
| 108 | | 7.3 Confidentiality and coding | 19 |
| 109 | | 7.4 Retention and destruction of project data and biological material | 20 |
| 110 | 8 | FUNDING / PUBLICATION / DECLARATION OF INTEREST | 20 |
| 111 | 9 | REFERENCES | 20 |
| 112 | | Appendix 1: Schedule of assessments | 1 |

113

# **GLOSSARY OF ABBREVATIONS**

115

| 116 | | |
|-----|--------|-------------------------------------------------------|
| 117 | AE | Adverse Event |
| 118 | BASEC | Business Administration System for Ethical Committees |
| 119 | BDI-II | Beck Depression Inventory - 2 |
| 120 | CRF | Case report form |
| 121 | FOPH | Federal Office of Public Health |
| 122 | HRA | Human Research Act |
| 123 | HRO | Ordinance on Human |
| 124 | NRS | Numeric rating scale |
| 125 | PI | Principal Investigator |
| 126 | SAE | Serious Adverse Event |
| 127 | SF-MPQ | Short form – McGill Pain Questionnaire |
| 128 | USB | University Hospital Basel |
| 129 | USZ | University Hospital Zurich |
| 130 | | |
| 131 | | |

Version 1.1, 02.05.2023

# 132 **STUDY SYNOPSIS**

| | Milhalm Dunan Doct |
|---|---|
| Sponsor / Sponsor- | Wilhelm Ruppen, Prof. |
| Investigator | Head of the Pain Unit |
| | Department of Anaesthesiology |
| | University Hospital of Basel (USB) |
| | Spitalstrasse 21 |
| | CH - 4031 Basel |
| | Phone: +41 61 328 64 96 |
| | Fax: +41 61 265 57 20 |
| | E-mail: wilhelm.ruppen@usb.ch |
| Study Title: | Lidocaine and ketamine levels in plasma after simultaneous lidocaine/ketamine infusions. An observational assessment of therapy effects and side-effects. |
| Short Title / Study ID: | LiKe-Level-Trial |
| | Version 1.1 (dated 02/05/2023) |
| Protocol Version and Date: | · · · |
| Trial registration: | The study will be registered at clinicaltrials.gov and the Swiss National clinical trial portal (SNCTP) upon ethical approval. |
| Study category and Rationale | Category A: Participants in this study will be exposed to minimal additional risks. |
| Background and | Around 20% of the European population suffers from chronic pain. In |
| Rationale: | addition to the huge emotional and physical burden of chronic pain, the |
| | financial impact on society is also enormous, currently estimated at more than €200 billion each year in Europe and \$150 billion each year in the USA. [1] However, there are many different treatment strategies for chronic pain, suggesting difficulties in effectively treating these patients. [2] In addition, a substantial number of patients do not respond to first-line treatment. [5] Medications that are frequently prescribed for pain (e.g., NSAIDs, acetaminophen, metamizole, opioids, antidepressants and antiepileptics) often have limiting side effects. [6] Opioids have the additional problem that they have a high potential for abuse and addiction. [7, 8] One possible treatment strategy, especially for therapy-resistant pain, is intravenous infusions with certain pharmacological agents, such as lidocaine and ketamine. [9] Studies have shown that treatments with lidocaine and ketamine have an immediate effect on the one hand, and can also result in longer-lasting pain relief on the other. [10-13] Lidocaine-ketamine infusions (every 4-6 weeks) have been performed at the University Hospital Basel (USB) for almost 20 years. In our pain unit, we combine the positive properties of lidocaine and ketamine by administering infusions of the two agents simultaneously. Internationally, however, safety concerns have been raised following some case studies reported serious side effects [17-19] and the death of a young mother reported in the British media after lidocaine infusion [20]. Therefore, in 2021, an international expert consensus was conducted on the efficacy and safety of intravenous lidocaine for postoperative pain. [21] The elaborated statement includes recommendations for the safe use of lidocaine infusions in the perioperative setting, such as: - A loading dose of no more than 1.5mg/kg lidocaine given as an intravenous infusion over 10 minutes is recommended - After the initial loading dose, an intravenous infusion of 1.5mg/kg/h lidocaine is recommended |

| Objective(s): | The dosage regimens proposed in this recommendation are clearly exceeded by the standard regime at our pain unit (i.e. 4mg/kg lidocaine over 30 minutes). For note the new consensus statement addresses perioperative use of lidocaine in acute postoperative pain, and our treatment regime is based on previous studies investigating chronic pain. [9, 22] In addition, during a previous retrospective study at our Pain Unit, no serious adverse events were registered during 2995 infusions performed, rendering it a safe procedure. [23] Nevertheless, Foo, Macfarlane et al. defined a toxic lidocaine concentration in plasma as >5µg/ml. In order to assess whether this concentration is exceeded at the USB, the aim of this pilot project is to measure the lidocaine plasma level in a limited number of patients to generate explorative data on inter- and intrapersonal stability and safety of drug plasma levels. Beyond safety issues, we are interested in dosing and effects of our treatments. In the literature, there is evidence that higher doses of ketamine are associated with greater and longer pain relief, which is also consistent with the data from our retrospective study. [23, 24] As a standard regime of our infusion therapies, we increase the ketamine dose from 0.15mg/kg at the first infusion to 0.25mg/kg at the second infusion and 0.5mg/kg at the third infusion. Therefore, another aim of this study is to investigate whether higher plasma levels of ketamine can be correlated with a better analgesic effect. The primary objective of this study is to measure the concentration of lidocaine in the plasma of patients at the USB after an intravenous infusion |
|---|---|
| | with 4mg/kg lidocaine over 30 minutes. We hypothesize that lidocaine concentrations in plasma of patients at the USB are inter- and intrapersonal stable and do not exceed 5µg/ml by the end of the applied infusions. |
| | The secondary objectives of this study include the prospective side effects assessment of lidocaine and ketamine as well as the measurement of plasma levels of ketamine. Further, to correlate the plasma levels with the analgesic efficacy and change in possible depressive symptoms, due to the infusions. |
| Outcome(s): | The primary endpoint of our study is the concentration of lidocaine in the plasma of patients who received an intravenous infusion with 4mg/kg lidocaine and 0.15 – 0.5mg/kg ketamine over 30 minutes at the time directly after the infusion. |
| | The secondary endpoints of our study are the recorded side-effects typical for lidocaine and ketamine reported by questionnaires and patient monitoring. A further endpoint of interest is the concentration of ketamine in the plasma of patients directly after the infusion. Development of pain and mood as assessed by the Short form - McGill Pain Questionnaire (SF-MPQ) and Beck Depression Questionnaire II (BDI-II), respectively. |
| Study design: | This study is designed as monocentric observational study at the University Hospital Basel. |

# Inclusion / Exclusion criteria:

#### Inclusion Criteria:

- Patient is a new recipient of lidocaine-ketamine infusions
- Patient is 18 years of age or older
- Patient is able to provide Informed Consent

#### **Exclusion Criteria:**

- Contraindication to blood sampling (on arm **not used** for infusion)
- Insufficient knowledge of German language
- Inability to give consent
- Patient is under 18 years of age
- Contraindication to treatment with lidocaine and/or ketamine

# Measurements and procedures:

# Standard procedure of lidocaine/ketamine infusions at USB

Patients with therapy refractory chronic pain are scheduled for Infusion therapies on a four-week interval basis, by their treating pain physician. Before each infusion, a brief medical history interview takes place, during which compliance with the fasting time (6 hours for solid food, 2 hours for clear liquids) in particular is queried. Subsequently, installation of monitoring (10-minute blood pressure measurement, continuous 5-lead ECG, and continuous SPO2 measurement) and placement of venous access. Lidocaine and ketamine are infused over a 30-minute period (detailed dosing schedules are provided in the protocol). After infusion, patients are monitored for at least another half hour, discharged in company, and instructed not to operate heavy machinery or motor vehicles for at least 24 hours. Over the first three infusions the Ketamine dose is adjusted up to 0.5mg/kg/bw, the Lidocaine dose is stable at 4mg/kg/bw during the infusions. Beyond the third infusion dose adjustments are only made if needed (c.f. side-effects)

#### Study procedures

Recruitment and consent to participate in the study will take place in the consultation prior to the first infusion. (c.f. 3.2) During the infusion, the patients' vital signs will be monitored as usual (10-minute blood pressure measurement, continuous SPO2 and 5-lead ECG are recorded, c.f. 3.3.2). As a part of this study, at the end of the first, second and third infusion, side effects will be screened using customized questionnaires. (c.f. eCRF forms document). In addition, blood will be collected during each of the first three infusion appointments. The blood collection itself will take place within 3 minutes after termination of the infusion, as we assume the highest plasma levels at that point in time. [25, 26] For blood collection we will use a Butterfly cannula (BBraun Venofix® Safety 23G, PZN 08839883, B. Braun Melsungen AG) which will be inserted on the "non-infusion arm" and two green 7.5ml Lithium-Heparin monovettes (S-Monovette® Lithium-Heparin, liquid, preparation: lithium heparin, liquid, 7.5 ml, membrane screw cap, closure green, color code ISO, (LxØ) without closure: 92 x 15 mm, with paper label, label/printing: green Sarstedt AG & Co. KG, Nümbrecht).

Patients will complete the Short form - McGill Pain Questionnaire (with additional recording of pain on the numeric rating scale (NRS) from 0 (no pain at all) to 10 (worst pain imaginable)) and Beck Depression Questionnaire directly prior to the first three infusions. The SF – MPQ is a validated instrument for measures of clinical pain that capture its sensory, affective and other qualitative components. [27] The BDI-II provides a validated psychological test procedure that assesses the severity of

depressive symptoms in adolescents 13 years of age and older and adults. [28]

In addition, these questionnaires will also be completed at the time points 7 days after, and 14 days after the first, second and third Infusion. The participants will receive a link by e-mail so that they can fill in the questionnaires online. According to the license agreement, the BDI-II will be filled out in paper form and the results will be subsequently transferred to REDCap. If desired by the participant, these questionnaires can also be completed during a telephone survey conducted by the study staff. The surveys will be conducted with REDCap. After the third infusion, this online questioning will take place additionally after 28 days (c.f. Appendix 1). After this questioning, the study ends for the participants.

### Investigated variables

#### **Demographic**

Variable: Age

Categories: Age at beginning of therapy (recorded in years)

Variable: Gender

Categories: female / male / diverse

Variable: Nationality

Categories: Recorded as free text

Variable: Diagnosis that led to the indication for lidocaine/ketamine

infusion

Categories: Main pain-related diagnosis coded with ICD11, free text

Variable: Dosage

Categories: Weight (recorded in kg) / Height (recorded in cm) / Dosage of lidocaine (recorded in mg) / Dosage of ketamine (recorded in mg)

#### **Effects and Side effects**

Variable: Depressive Symptoms

Categories: Recorded by BDI-II at the beginning of the infusion, 7 days

after and 14 days after

Variable: Pain

Categories: Recorded by SF-MPQ-2 at the beginning of the infusion, 7 days after and 14 days after, and by NRS (Number from 0 to 10) at the beginning of the infusion, 7 days after and 14 days after

Variable: Vital sings

Categories: blood pressure (recorded in mmHg) / heart rate (recorded in bpm) / saturation of oxygen under infusion (recorded as percentage) / Respiratory rate (recorded in breaths per minute), recorded at the start of the infusion and subsequently during a period of 60 minutes

Variable: ECG

Categories: Heart rate (recorded in bpm), regular sinus rhythm (recorded as yes or no), PQ interval (recorded in ms), QRS-complex (recorded in ms), ST segment (recorded as conspicuous/inconspicuous), T wave (recorded as conspicuous/inconspicuous), QTc (recorded in ms), Extrasystolies (recorded as number), other anomalies (recorded as free text) at start of infusion and at the end of infusion (minute 30)

Variable: Side effects at end of infusion (patient recorded)

| | Categories: Injection site pain, dysphoria, euphoria, nervousness, anxiety, dyspnea, nausea, hypersalivation, nightmares, hallucinations, visual disturbances, tinnitus, hyperacusis, paresthesias, numbness, dizziness (recorded as present/absent). |
|---|---|
| | Variable: Side effects at end of infusion (patient observation by physician, monitoring) Categories: Exanthema, redness injection site, vomiting, tremor, dysarthria, nystagmus, convulsions, dissociation, disorientation, restlessness, agitation (recorded as present/absent) |
| | Variable: Medication plasma levels Categories: Lidocaine and ketamine plasma levels are recorded specified in mg/l al the end of infusions |
| | Laboratory Analysis |
| | Samples were analyzed on a Thermo Scientific™ Orbitrap Exploris™ 240 Mass Spectrometer coupled to reversed phase liquid chromatography with an LLOQ of 0.1 µmol/L for lidocaine and 0.1 mg/L for ketamine. The methods were fully validated according to EMA guideline. |
| Number of<br>Participants with<br>Rationale: | A total of max. 15 patients (10 + Drop-out of 50%) will be included. |
| Study Duration: | In total, we expect a study duration of 7 months. Study duration for each individual participant will be 12 weeks. |
| Study Schedule: | First-Participant-In: 06/2023 Last-Participant-Out: 12/2023 |
| Principal Investigator and Project Leader: | Wilhelm Ruppen, Prof. Leiter der Schmerzklinik Klinik für Anästhesiologie |
| | Universitätsspital Basel (USB) |
| | Spitalstrasse 21 |
| | CH - 4031 Basel |
| | Telefon: +41 61 328 64 96<br>Fax: +41 61 265 57 20 |
| | E-mail: wilhelm.ruppen@usb.ch |
| | Tobias Schneider, MD |
| | Senior Physician |
| | Department of Anaesthesiology |
| | University Hospital of Basel (USB) Spitalstrasse 21 |
| | CH - 4031 Basel |
| | Phone: +41 61 328 65 43 |
| | Phone: +41 61 328 65 43 Fax: +41 61 265 57 20 E-mail: tobias.schneider@usb.ch |

### Co-Investigator(s):

Flavia Flepp, pract. med.

Doctoral candidate

Department of Anaesthesiology University Hospital of Basel (USB)

Spitalstrasse 21 CH - 4031 Basel

Phone: +41 61 556 55 73 Fax: +41 61 265 57 20

E-mail: flaviabarla.flepp@usb.ch

Matthijs de Leeuw, pract. med.

Doctoral candidate

Department of Anaesthesiology University Hospital of Basel (USB)

Spitalstrasse 21 CH - 4031 Basel

Phone: +41 61 328 59 14 Fax: +41 61 265 57 20

E-mail: matthijsjan.deleeuw@usb.ch

Regula Steiner, Dr. sc. nat.

Head of Laboratory for Therapeutic Drug Monitoring and Toxicology

Institute for Clinical Chemistry University Hospital of Zurich (USZ)

OPS D29

Rämistrasse 100 CH - 8091 Zurich

Phone: +41 43 253 06 09 E-mail: regula.steiner@usz.ch

### Study Centre(s):

University Hospital of Basel (USB)

Spitalstrasse 21 CH - 4031 Basel

# Statistical Considerations:

Patients characteristics regarding to age, gender, pharmacological treatment, medical diagnosis will be analyzed exploratively/ descriptively.

#### **Primary outcome:**

The primary outcome (Lidocaine plasma level) of our study is explorative and not comparative, therefore, no H0 or H1 are formulated no power analysis is performed and only descriptive/ explorative statistics are reported.

We plan to include 10 patients with complete data sets, meaning, full data of three infusions with stable dose of lidocaine (4mg/kg/BW) and escalating dose of ketamine (0.15 – 0.5mg/kg/BW). This corresponds to thirty measures of lidocaine plasma concentrations at a dose of 4mg/kg/BW). Patients without full data sets will be replaced but data from patients with preliminary study termination will be reported in the final protocol.

## **Secondary outcomes:**

- 1. Ketamine plasma levels are assessed according to lidocaine levels.
- 2. H0: dose escalation of ketamine has no effect on pain (outcome measure: SF-MPQ-2) and mood (outcome measure: BDI-II. H1: we hypothesize that ketamine dose has an effect on both outcome measures. For repeated measurements, an ANOVA will be separately calculated for outcome measures of pain and mood as dependent variable. This analysis will be performed separately for intermediate (one and two weeks) and

| | significance of 0.05 will be used. In case of multiple testing a correction factor (in case of ANOVA: Bonferroni) for multiple testing is applied. 3. Side effects during treatment will be primary analyzed descriptively. |
|---|---|
| | 4. Multiple exploratory linear regressions will be calculated to evaluate the impact of dose and plasma levels of lidocaine and ketamine on pain and mood as well as occurrence of side-effects. |
| | SPSS Version 25 will be used for data analyzation and graph pad PRISM Version 9 for data visualization. The investigators, Flavia Flepp and Tobias Schneider, will perform all analysis steps. If needed, statistical guidance will be applied by statisticians of the Clinical Trial Unit (CTU) of the USB. |
| | Handling of missing data: |
| | Dropouts will be replaced. We do not plan data imputation. |
| GCP Statement: | This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements. |

135

136

137

138

139

140

141

142143

144

145

146

147

148

149

150

151 152

153

154

155

156

157158

### 1 BACKGROUND AND PROJECT RATIONALE

Around 20% of the European population suffers from chronic pain. In addition to the huge emotional and physical burden of chronic pain the financial impact on society is also enormous, currently estimated at more than €200 billion each year in Europe and \$150 billion each year in the USA. [1] Moreover, chronic pain is the most common cause of long-term disability in middleaged people. [2] Chronic pain is complex and the pathomechanisms behind it are still not fully understood. Nevertheless, it is increasingly regarded not only as a symptom, but as a disease in its own right. This is also visible in the fact that chronic pain can be coded independently for the first time in ICD 11. [3] In recent years, clinical research has shown that chronic pain can occur independently of disease or tissue damage due to increased sensitization of the central or peripheral nervous system. If chronic pain is inadequately treated, it leads to multidimensional adverse effects: Impairments in daily activities and work ability, general health, and social life. [4] However, there are many different treatment strategies for chronic pain, suggesting difficulties in effectively treating these patients. [2] In addition, a substantial number of patients do not respond to first-line treatment. [5] Medications that are frequently prescribed for pain (e.g., NSAIDs, acetaminophen, metamizole, opioids, antidepressants and antiepileptics) often have limiting side effects. [6] Opioids have the additional problem that they have a high potential for abuse and addiction. [7, 8]

One possible treatment strategy, especially for therapy-resistant pain, is intravenous infusions with certain pharmacological agents, such as lidocaine and ketamine [9] Studies have shown that treatments with lidocaine and ketamine have an immediate effect on the one hand, and can also result in longer-lasting pain relief on the other. [10-13] Ketamine is also interesting for pain therapy due to its antidepressant effect [14, 15] since chronic pain is often accompanied by depressive symptoms. [16]

Lidocaine-ketamine infusions (every 4-6 weeks) have been performed at the University Hospital Basel (USB) for almost 20 years. In our pain unit, we combine the positive properties of lidocaine and ketamine by administering infusions of the two agents simultaneously. This allows us to achieve good clinical results in patients who are non-responders to first- or second-line therapy. Internationally, however, safety concerns have been raised following some case studies reported serious side effects [17-19] and the death of a young mother reported in the British media after lidocaine infusion. [20] Therefore, in 2021, an international expert consensus was conducted on the efficacy and safety of intravenous lidocaine for postoperative pain. [21] The elaborated statement includes recommendations for the safe use of lidocaine infusions in the perioperative setting, such as:

- 170 A loading dose of no more than 1.5mg/kg lidocaine given as an intravenous infusion over 10 minutes is recommended
  - After the initial loading dose, an intravenous infusion of 1.5mg/kg/h lidocaine is recommended
    - No more than 120mg/h of lidocaine should be infused intravenously
  - For the dose calculation, the ideal body weight should be used

The dosage regimens proposed in this recommendation are clearly exceeded by the standard regime at our pain unit (i.e. 4mg/kg lidocaine over 30 minutes). For note the new consensus statement addresses perioperative use of lidocaine in acute postoperative pain, and our treatment regime is based on previous studies investigating chronic pain. [9, 22] In addition, during a previous retrospective study at our Pain Unit, no serious adverse events were registered during 2995 infusions performed, rendering it a safe procedure. [23] Nevertheless, Foo, Macfarlane et al. defined a toxic lidocaine concentration in plasma as >5µg/ml. In order to assess whether this concentration is exceeded at the USB, the aim of this pilot project is to measure the lidocaine plasma level in a limited number of patients to generate explorative data on inter- and intrapersonal stability and safety of drug plasma levels.

Beyond safety issues, we are interested in dosing and effects of our treatments. In the literature, there is evidence that higher doses of ketamine are associated with greater and longer pain relief, which is also consistent with the data from our retrospective study. [23, 24] As a standard regime of our infusion therapies, we increase the ketamine dose from 0.15mg/kg at the first infusion to 0.25mg/kg at the second infusion and 0.5mg/kg at the third infusion. In cases where patients already experiencing sufficient analgesic effect and/or improvement in quality of life after the 1st or 2nd infusion or if side effects are not tolerated, no further increase of ketamine dosage is made. Therefore, another aim of this study is to investigate whether higher plasma levels of ketamine can be correlated with a better analgesic effect.

# 2 PROJECT OBJECTIVES AND DESIGN

# 2.1 Hypothesis and primary objective

- The primary objective of this study is to measure the concentration of lidocaine in the plasma of patients at the USB after an intravenous infusion with 4mg/kg lidocaine over 30 minutes.
- We hypothesize that lidocaine concentrations in plasma of patients at the USB are inter- and intrapersonal stable and do not exceed 5µg/ml by the end of the applied infusions.

# 2.1.2 Secondary objectives

The secondary objectives of this study include the prospective side effects assessment of lidocaine and ketamine as well as the measurement of plasma levels of ketamine. Further, to correlate the plasma levels with the analgesic efficacy and change in possible depressive symptoms, due to the infusions.

### 2.2 Primary and secondary endpoints

The primary endpoint of our study is the concentration of lidocaine in the plasma of patients who received an intravenous infusion with 4mg/kg lidocaine and 0.15 – 0.5mg/kg ketamine over 30 minutes at the time directly after the infusion.

The secondary endpoints of our study are the recorded side-effects typical for lidocaine and ketamine reported by questionnaires and patient monitoring. A further endpoint of interest is the concentration of ketamine in the plasma of patients directly after the infusion. Development of pain and mood as assessed by the Short form - McGill Pain Questionnaire (SF-MPQ) and Beck Depression Questionnaire II (BDI-II), respectively.

# 2.3 Project design

This study is designed as monocentric observational pilot-study at the USB.



# 3 PROJECT POPULATION AND STUDY PROCEDURES

### 3.1 Project population, inclusion and exclusion criteria

For our pilot project on drug plasma levels in an ambulatory infusion regime, a total of max. 15 patients (10 + Drop-out of 50%) newly receiving lidocaine-ketamine infusions at the USB will be randomly selected. To minimize selection bias (including only responders, or patients with less side-effects) and because we increase the ketamine dosage normally during the first 3 infusions, we will only include patients who are new to lidocaine/ketamine infusions.

#### Inclusion Criteria:

- Patient is a new recipient of lidocaine-ketamine infusions

- 234 - Patient is 18 years of age or older
- 235 - Patient is able to provide Informed Consent

- 237 **Exclusion Criteria:**
- 238 - Contraindication to blood sampling (on arm not used for infusion)
- 239 - Insufficient knowledge of German language
- 240 - Inability to give consent
- 241 - Patient is under 18 years of age
- 242 - Contraindication to treatment with lidocaine and/or ketamine

243

#### 244 3.2 Recruitment, screening and informed consent procedure

- 245 All patients who are newly assigned to lidocaine-ketamine infusions at the USB and who meet
- 246 the inclusion criteria will be asked to take part in the study by their treating physician.
- 247 If the patients are willing to participate, they will be informed in verbal and written form by one of
- 248 the investigators about the study and the blood collection.
- 249 All study participants will receive an informed consent form describing the study and providing
- 250 sufficient information to allow participants to make an informed decision about their participation
- 251 in the study. Sufficient time (at least 24 hours) will be given to the potential participants to make
- 252 a decision about participation.
- 253 Formal informed consent will be obtained from a participant using the approved consent form
- 254 before the participant undergoes any of the study procedures.
- 255 The consent form will be signed and dated by the investigator or his/her designee concurrently
- 256 with the participant's signature. A copy of the signed consent form will be given to the study
- 257 participant. The informed consent form will be retained as part of the study records.
- 258 The patients themselves have no direct advantage from participating in the study. The risk
- 259 resulting from an additional venepuncture is to be considered minimal. The typical risks of
- 260 inserting an indwelling venous cannula are already part of the infusion information. However,
- 261 patients are explicitly informed that taking part in the study includes three additional venous
- 262 punctures.

263

# 3.3 Study procedures

- 264 Recruitment and consent to participate in the study will take place in the consultation prior to the
- 265 first infusion. (c.f. 3.2) During the infusion, the patients' vital signs will be monitored as usual (10-
- 266 minute blood pressure measurement, continuous SPO2 and 5-lead ECG are recorded, c.f. 3.3.2).
- 267 As a part of this study, at the end of the first, second and third infusion, side effects will be
- 268 screened using customized questionnaires (c.f. eCRF forms document). In addition, blood will be
- 269 collected during each of the first three infusion appointments. The blood collection itself will take
- place within 3 minutes after termination of the infusion, as we assume the highest plasma levels 270
- 271 at that point in time. [25, 26] For blood collection we will use a Butterfly cannula (BBraun Venofix®
- 272 Safety 23G, PZN 08839883, B. Braun Melsungen AG) which will be inserted on the "non-infusion
- 273 arm" and two green 7.5ml Lithium-Heparin monovettes (S-Monovette® Lithium-Heparin liquid, 274 preparation: lithium heparin, liquid, 7.5 ml, membrane screw cap, closure green, color code ISO,
- 275 (LxØ) without closure: 92 x 15 mm, with paper label, label/printing: green Sarstedt AG & Co. KG,
- Nümbrecht). 276
- 277 Patients will complete the Short form - McGill Pain Questionnaire (with additional recording of
- 278 pain on the numeric rating scale (NRS) from 0 (no pain at all) to 10 (worst pain imaginable)) and
- 279 Beck Depression Questionnaire directly prior to the first three infusions. The SF - MPQ is a
- 280 validated instrument for measures of clinical pain that capture its sensory, affective and other

- 281 qualitative components. [27] The BDI-II provides a validated psychological test procedure that
- 282 assesses the severity of depressive symptoms in adolescents 13 years of age and older and
- 283 adults. [28]
- 284 In addition, these questionnaires will also be completed at the time points 7 days after, and 14
- 285 days after the first, second and third Infusion. The participants will receive a link by e-mail so that
- 286 they can fill in the questionnaires online. According to the license agreement, the BDI-II will be
- 287 filled out in paper form and the results will be subsequently transferred to REDCap. If desired by
- 288 the participant, these questionnaires can also be completed during a telephone survey conducted
- by the study staff. The surveys will be conducted with REDCap. After the third infusion, this online 289
- 290 questioning will take place additionally after 28 days (c.f. Appendix 1). After this questioning, the
- 291 study ends for the participants.

293

## 3.3.1 Investigated variables

294 295

# **Demographic**

296

- 297 Variable: Age
- 298 Categories: Age at beginning of therapy (recorded in years)

299

- 300 Variable: Gender
- 301 Categories: female / male / diverse

302

- 303 Variable: Nationality
- 304 Categories: Recorded as free text

305

- 306 Variable: Diagnosis that led to the indication for lidocaine/ketamine infusion
- 307 Categories: Main pain-related diagnosis coded with ICD11, free text
- 308 Variable: Dosage
- 309 Categories: Weight (recorded in kg) / Height (recorded in cm) / Dosage of lidocaine (recorded in
- 310 mg) / Dosage of ketamine (recorded in mg)

#### 311 **Effects and Side effects**

- 312 Variable: Depressive Symptoms
- 313 Categories: Recorded by BDI-II at the beginning of the infusion, 7 days after and 14 days after
- 314 Variable: Pain
- 315 Categories: Recorded by SF-MPQ-2 at the beginning of the infusion, 7 days after and 14 days
- 316 after, and by NRS (Number from 0 to 10) at the beginning of the infusion, 7 days after and 14
- 317 days after
- 318 Variable: Vital sings
- 319 Categories: blood pressure (recorded in mmHg) / heart rate (recorded in bpm) / saturation of
- 320 oxygen under infusion (recorded as percentage) / Respiratory rate (recorded in breaths per
- 321 minute), recorded at the start of the infusion and subsequently during a period of 60 minutes
- 322 Variable: ECG
- 323 Categories: Heart rate (recorded in bpm), regular sinus rhythm (recorded as yes or no), PQ
- 324 interval (recorded in ms), QRS-complex (recorded in ms), ST segment (recorded as
- 325 conspicuous/inconspicuous), T wave (recorded as conspicuous/inconspicuous), QTc (recorded
- 326 in ms), Extrasystolies (recorded as number), other anomalies (recorded as free text) at start of
- 327 infusion and at the end of infusion (minute 30)

- 328 Variable: Side effects at end of infusion (patient recorded)
- 329 Categories: Injection site pain, dysphoria, euphoria, nervousness, anxiety, dyspnea, nausea,
- hypersalivation, nightmares, hallucinations, visual disturbances, tinnitus, hyperacusis,
- paresthesias, numbness, dizziness (recorded as present/absent).
- Variable: Side effects at end of infusion (patient observation by physician, monitoring)
- Categories: Exanthema, redness injection site, vomiting, tremor, dysarthria, nystagmus,
- convulsions, dissociation, disorientation, restlessness, agitation (recorded as present/absent)

- 336 Variable: Medication plasma levels
- Categories: Lidocaine and ketamine plasma levels are recorded specified in mg/l al the end of
- 338 infusions

### 3.3.2 Standard Procedure of lidocaine-ketamine infusions at the Pain Unit of USB

339340

- During a short medical history interview Patients are briefly asked about their current pain situation before each infusion. For safety reasons, additional questions are asked about weight changes, compliance with fasting (= no solid food for 6 hours, no drinks for 2 hours) and allergies.
- Monitoring is then installed (10-minute blood pressure measurement, continuous SPO2 and 5-lead ECG are recorded) and venous access is established. Lidocaine and ketamine are infused
- over a period of 30 minutes. The dosage of lidocaine is 4mg/kg is maintained throughout the infusions, and the dosage of ketamine is increased within the first three infusions from 0.15mg/kg.
- infusions, and the dosage of ketamine is increased within the first three infusions from 0.15mg/kg at the first, to 0.25mg/kg at the second and 0.5mg/kg at the third infusion. In case patients already
- experiencing sufficient analgesic effect and/or improvement in quality of life after the 1st or 2nd
- infusion or if side effects do not allow a further dose increase, no further step up of ketamine
- dosage is made. We define a sufficient effect as a significant pain reduction (more than 50%) for at least 2 weeks and/or better quality of life with improved functionality during at least 2 weeks.
- After the infusion, patients are monitored for at least another half hour, are discharged in company and are instructed to not run heavy machines and motor vehicles for at least 24 hours.

355356

### 3.3.3 Laboratory Analysis

- Plasma concentrations of lidocaine and ketamine are determined at the Institute of clinical chemistry at University Hospital Zurich under ISO/IEC 17025:2017 accreditation.
- The Plasma lidocaine and ketamine concentrations are measured using liquid chromatography coupled to high-resolution accurate mass-spectrometry (LC-MS).
- For lidocaine measurement, 100uL of plasma samples are precipitated with 100uL acetonitrile (containing internal standard) and centrifuged. Supernatant is diluted with 5mM ammonium format
- 363 buffer pH 3 for analysis.
- For ketamine measurement, 1 mL of plasma samples are diluted with 0.5mL H2O and 0.5 mL
- ethanol (containing internal standard) extracted using e 150 µl 1 M NaOH in H2O and 5 ml n-
- Hexan/Dichlormethan (4+1, v+v). Supernatant was separated and dried down under steam of N2.
- For measurement, samples are reconstituted with acetonitrile and 10 mM ammonium acetate
- 368 buffer.
- 369 Samples were analyzed on a Thermo Scientific™ Orbitrap Exploris™ 240 Mass Spectrometer
- 370 coupled to reversed phase liquid chromatography with an LLOQ of 0.1 µmol/L for lidocaine and
- 371 0.1 mg/L for ketamine. The methods were fully validated according to EMA guideline.
- Both methods were fully validated according to EMA guideline.

373

374

#### 3.4 Withdrawal and discontinuation

Patients may withdraw from the study at any time and for any reason (stating reason is not

- required). No further data will be collected after withdrawal. Unless otherwise requested, the data collected up to that point will still be evaluated in encrypted form and anonymized after the evaluation.
- 379 The following reasons result in withdrawal:
- 380 SAE
  - AE challenging the health of the subject if continuing the study

Drop-outs will be replaced by new patients and will be reported in the final publication.

# 384

385

386

381

382

## 4 STATISTICS AND METHODOLOGY

# 4.1. Statistical analysis plan

Patients characteristics regarding to age, gender, pharmacological treatment, medical diagnosis will be analyzed exploratively/ descriptively.

# 389 390

# Primary outcome:

- The primary outcome (Lidocaine plasma level) of our study is explorative and not comparative, therefore no H0 or H1 are formulated no power analysis is performed and only descriptive/ explorative statistics are reported.
- We plan to include 10 patients with complete data sets, meaning, full data of three infusions with stable dose of lidocaine (4mg/kg/BW) and escalating dose of ketamine (0.15 0.5mg/kg/BW). This corresponds to thirty measures of lidocaine plasma concentrations at a dose of 4mg/kg/BW).
- Patients without full data sets will be replaced but data from patients with preliminary study termination will be reported in the final protocol.

# 399 400

## Secondary outcomes:

1. Ketamine plasma levels are assessed according to lidocaine levels.

401 402 403

404

405

406 407

408

2. H0: dose escalation of ketamine has no effect on pain (outcome measure: SF-MPQ-2) and mood (outcome measure: BDI-II. H1: we hypothesize that ketamine dose has an effect on both outcome measures. For repeated measurements, an ANOVA will be separately calculated for outcome measures of pain and mood as dependent variable. This analysis will be performed separately for intermediate (one and two weeks) and long term effects (four weeks). For comparative outcomes a level of significance of 0.05 will be used. In case of multiple testing, a correction factor (in case of ANOVA: Bonferroni) for multiple testing is applied.

409 410

3. Side effects during treatment will be primary analyzed descriptively.

411412413

4. Multiple exploratory linear regressions will be calculated to evaluate the impact of dose and plasma levels of lidocaine and ketamine on pain and mood as well as occurrence of side-effects.

414 415

420

- SPSS Version 25 will be used for data analyzation and graph pad PRISM Version 9 for data
- visualization. The investigators, Flavia Flepp and Tobias Schneider, will perform all analysis
- steps. If needed, statistical guidance will be applied by statisticians of the Clinical Trial Unit (CTU)

#### 419 of the USB.

## 4.2. Handling of missing data

Dropouts will be replaced (c.f. 3.4). We do not plan data imputation.

# 422 5 REGULATORY ASPECTS AND SAFETY

# 423 **5.1 Local regulations / Declaration of Helsinki**

- 424 This research project will be conducted in accordance with the protocol, the Declaration of
- Helsinki [3], the principles of Good Clinical Practice, the Human Research Act (HRA) and the
- Human Research Ordinance (HRO) [1] as well as other locally relevant regulations. The project
- leader acknowledges his responsibilities as both the project leader and the Sponsor.

# 428 5.2 Notification of safety and protective measures (HRA Art. 15, HRO Art. 20)

- 429 If, during the research project, circumstances arise which could jeopardise the safety or health of
- 430 the participants or lead to a disproportionate relationship between the risks and burdens and the
- benefits, all the measures required to ensure protection are to be taken without delay.
- The project leader is promptly notified (within 24 hours) if immediate safety and protective
- 433 measures have to be taken during the conduct of the research project. The Ethics Committee will
- be notified via BASEC of these measures and of the circumstances necessitating them within 7
- 435 days.

# 436 **5.3 Serious events (HRO Art. 21)**

- 437 If a serious event occurs, the research project will be interrupted and the Ethics Committee
- notified on the circumstances via BASEC within 7 days according to HRO Art. 21<sup>1</sup>.

#### 439 **5.4 Amendments**

- Substantial changes to the project set-up, the protocol and relevant project documents will be
- submitted to the Ethics Committee for approval according to HRO Art. 18 before implementation.

# **442 5.5** End of project

- 443 Upon project completion or discontinuation, the Ethics Committee is notified within 90 days. All
- biological materials and health-related data are anonymized upon termination of data analysis.

### **5.6 Insurance**

- In the event of project-related damage or injuries, the Sponsor will be liable, except for damages
- 447 that are only slight and temporary; and for which the extent of the damage is no greater than
- could be expected according to the current state of scientific knowledge (Art. 12 HRO).

### 449 6 FURTHER ASPECTS

## 450 **6.1 Overall ethical considerations**

- Overall, this project is in accordance with the regulatory requirements of the HFG and the HFV.
- 452 An approval of the local ethic committee is mandatory to conduct this project. The minimal

<sup>&</sup>lt;sup>1</sup> A serious event is defined as any adverse event where it cannot be excluded, that the event is attributable to the sampling of biological material or the collection of health-related personal data, and which:

a. requires inpatient treatment not envisaged in the protocol or extends a current hospital stay;

b. results in permanent or significant incapacity or disability; or

c. is life-threatening or results in death.

- additional risks of an additional venous cannulation for the single patient is outweighed by far due
- 454 to the additional knowledge we generate about the safety profile and dose adjustments for
- patients receiving future infusion treatments. As this is an observational study and the blood
- sample analysis only evaluates the drug plasma levels, we do not expect incidental findings due
- 457 to study procedures. Especially the screening for depression is a standard procedure at the pain
- 458 clinics, suspicion of depression would be communicated to the patient independently of study
- participation. This is also the case for incidental findings during the hemodynamic monitoring
- 460 during the infusion therenice
- during the infusion therapies.

#### 6.2 Risk-Benefit Assessment

- Venous catherization brings the risk of bleeding, bruises, swellings with it, as well as the small
- 463 chance of infection.
- In summary, this study will not provide any direct benefit beyond the expected relief by the infusion
- therapy on pain, to the participating patients, but it may provide valuable insights as a basis from
- 466 which we can optimize and adopt our infusion regimes up on plasma levels of lidocaine and
- 467 ketamine correlated with effects and side-effects. Participants will be exposed to minimal
- additional risks due to the venous cannulation.

## 7 QUALITY CONTROL AND DATA PROTECTION

# 7.1 Quality measures

- The study will be conducted by a small team of the Pain Unit of the USB. All team members will
- be trained on all important study related aspects.
- 473 For quality assurance the sponsor, the Ethics Committee or an independent trial monitor may visit
- 474 the research sites. Direct access to the source data and all study related files is granted on such
- occasions. All involved parties keep the participant data strictly confidential.

476

477

469

470

461

## 7.2 Data recording and source data

- 478 Study data will be recorded with electronic CRFs, using a database (RedCap, Research
- 479 Electronic Data Capture, Vanderbilt University, Tennessee, USA). For each enrolled study
- participant CRFs will be maintained. Participants will not be identified in the CRF by name or
- initials and birth date; instead the participant number will be used. The study staff and the PIs are
- 482 authorized for all CRFs.
- 483 Demographic data, visit dates, participation in study and Informed Consent Forms, randomization
- 484 number, SAEs, AEs and concomitant medication, results of relevant examinations and all CRFs
- are considered the source documents in the study.
- Paper source documents will be archived in folders at the study site with restricted access (Pain
- 487 Unit USB).

488

489

# 7.3 Confidentiality and coding

- 490 Project data will be handled with uttermost discretion and is only accessible to authorized
- 491 personnel who require the data to fulfil their duties within the scope of the research project. On
- 492 the CRFs and other project specific documents, participants are only identified by a unique
- 493 participant number.
- The data collection is based on electronic CRFs, other source documents will be on paper. Data
- from paper forms will then be transferred to the source documentation in a secure database. Only
- 496 Cls and study team members will be authorized to coordinate CRF entries. Data entry of paper

- pencil documents will be checked double after entry into the eCRF. The electronic database is based on the secure web application REDCap (Research Electronic Data Capture) and will be operated with individual user log in, time stamp, and logging of changes with the name of the respective study member. Only authorized personnel will be able to enter the system to view and edit data.
- Participants will not be identified in the CRF by name or initials and birth date. Only participant identification codes will be used to track participants. The participant identification list will be stored at the Pain Unit and will be only accessible for the investigators. The data will be locked and therefore protected from unauthorized or accidental disclosure, alteration, deletion, copying and theft.

Biological material in this project is not identified by participant name but by a unique participant number. Biological material is appropriately stored in a restricted area only accessible to authorized personnel. The plasma samples analyzed by the laboratory of the USZ are coded with a unique batch and no personal/ identifying data will be shared with the USZ. The identification list is stored locked and protected from unauthorized access at the Pain Unit USB.

# 513 7.4 Retention and destruction of project data and biological material

- All study data will be archived for a minimum of 10 years after study termination or premature termination of the clinical trial. All data is archived in folders at the study site with restricted access (Pain unit USB).
- 517 Upon conclusion, the database is secured and cannot be changed anymore. The Plasma samples will be disposed by the laboratory of the USZ directly after analysis.

# 8 FUNDING / PUBLICATION / DECLARATION OF INTEREST

521 The study is funded by the Clinic for Anesthesia, USB. There is no conflict of interest and the 522 financing party has no influence on the protocol, analysis or publication. We plan to publish the 523 results in a peer-reviewed scientific journal. Upon request, we will provide the full study protocol 524 and data (as required by some journals). The trial results might be presented at scientific 525 congresses. The main publication will be created by Flavia Flepp, Matthijs de Leeuw, Regula 526 Steiner, Tobias Schneider and Wilhelm Ruppen. No unpublished data may be transmitted to a 527 third party without prior written approval by sponsors and PIs. No publication or communication 528 involving the results of the study is authorized without prior written consent from the PIs. In view 529 of patent and confidentiality issues, however, the PIs must accept requirements on the timing of 530 early publication. No use of professional writers is intended. The PIs will have ultimate authority 531 over any of the activities.

# 9 REFERENCES

507

519

520

- van Hecke, O., N. Torrance, and B.H. Smith, *Chronic pain epidemiology and its clinical relevance.* Br J Anaesth, 2013. **111**(1): p. 13-8.
- Scascighini, L., et al., *Multidisciplinary treatment for chronic pain: a systematic review of interventions and outcomes.* Rheumatology (Oxford), 2008. **47**(5): p. 670-8.
- 537 3. WHO. *ICD-11*. 2019 [cited 2023 15.03.]; Available from: 538 http://id.who.int/icd/entity/1581976053
- 539 4. Clauw, D.J., et al., *Reframing chronic pain as a disease, not a symptom: rationale and implications for pain management.* Postgrad Med, 2019. **131**(3): p. 185-198.

- 541 5. Norbury, A. and B. Seymour, Response heterogeneity: Challenges for personalised medicine and big data approaches in psychiatry and chronic pain. F1000Res, 2018. **7**: p. 55.
- 544 6. Coles, S., W. Dabbs, and S. Wild, *Pharmacologic Management of Chronic Pain.* Prim Care, 2022. **49**(3): p. 387-401.
- 546 7. Blondell, R.D., M. Azadfard, and A.M. Wisniewski, *Pharmacologic therapy for acute pain.* Am Fam Physician, 2013. **87**(11): p. 766-72.
- 548 8. Cohen, S.P., L. Vase, and W.M. Hooten, *Chronic pain: an update on burden, best practices, and new advances.* Lancet, 2021. **397**(10289): p. 2082-2097.
- 550 9. Kosharskyy, B., et al., *Intravenous infusions in chronic pain management.* Pain Physician, 2013. **16**(3): p. 231-49.
- 552 10. Niesters, M., C. Martini, and A. Dahan, *Ketamine for chronic pain: risks and benefits.* Br J Clin Pharmacol, 2014. **77**(2): p. 357-67.
- Horvat, S., B. Staffhorst, and J.M.G. Cobben, *Intravenous Lidocaine for Treatment of Chronic Pain: A Retrospective Cohort Study.* J Pain Res, 2022. **15**: p. 3459-3467.
- Tran, K. and S. McCormack, CADTH Rapid Response Reports, in Ketamine for Chronic
   Non-Cancer Pain: A Review of Clinical Effectiveness, Cost-Effectiveness, and Guidelines.
   2020, Canadian Agency for Drugs and Technologies in Health
- 559 Copyright © 2020 Canadian Agency for Drugs and Technologies in Health.: Ottawa (ON).
- Tully, J., et al., *Utilization of Intravenous Lidocaine Infusion for the Treatment of Refractory Chronic Pain.* Anesth Pain Med, 2020. **10**(6): p. e112290.
- 562 14. Jelen, L.A. and J.M. Stone, *Ketamine for depression.* Int Rev Psychiatry, 2021. **33**(3): p. 207-228.
- 564 15. McIntyre, R.S., et al., *Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation.* Am J Psychiatry, 2021. **178**(5): p. 383-399.
- 567 16. Goesling, J., L.A. Lin, and D.J. Clauw, *Psychiatry and Pain Management: at the Intersection of Chronic Pain and Mental Health.* Curr Psychiatry Rep, 2018. **20**(2): p. 12.
- 570 17. Afacan, M.A., et al., *Lidocaine-induced delirium: a case report.* Am J Emerg Med, 2015. 571 33(4): p. 603.e1-2.
- 572 18. Daraz, Y.M. and O.H. Abdelghffar, *Lidocaine Infusion: An Antiarrhythmic With Neurologic Toxicities.* Cureus, 2022. **14**(3): p. e23310.
- 574 19. Digala, L.P. and S. Lucchese, *IV Lidocaine Infusion Leading to the Toxic Levels in Serum Causing Asystole A Case Report.* Headache, 2020. **60**(1): p. 269-270.
- 576 20. Warburton, D. *Mum dies after two heart attacks when hospital gave her unlicensed drugs*. The Mirror 2019; Available from: <a href="https://www.mirror.co.uk/news/uk-news/mum-dies-after-two-heart-21100201">https://www.mirror.co.uk/news/uk-news/mum-dies-after-two-heart-21100201</a>
- Foo, I., et al., *The use of intravenous lidocaine for postoperative pain and recovery: international consensus statement on efficacy and safety.* Anaesthesia, 2021. **76**(2): p.
  238-250.
- Tremont-Lukats, I.W., et al., *Systemic administration of local anesthetics to relieve* neuropathic pain: a systematic review and meta-analysis. Anesth Analg, 2005. **101**(6): p. 1738-1749.
- 585 23. Striebel, J., T. Schneider, and W. Ruppen, Simultaneous Application of Lidocaine and Ketamine During an Ambulatory Infusion Therapy as a Treatment Option in Refractory Chronic Pain Conditions A retrospective analysis, in Pain Unit, Clinic for Anaesthesiology University Hospital Basel. 2022. Unpublished data under review.

- 589 24. Orhurhu, V., et al., *Ketamine Infusions for Chronic Pain: A Systematic Review and Meta-analysis of Randomized Controlled Trials.* Anesth Analg, 2019. **129**(1): p. 241-254.
- 591 25. Berk, T. and S.D. Silberstein, *The Use and Method of Action of Intravenous Lidocaine* and *Its Metabolite in Headache Disorders.* Headache, 2018. **58**(5): p. 783-789.
- Weinberg, L., et al., *Pharmacokinetics and pharmacodynamics of lignocaine: A review.*World Journal of Anesthesiology, 2015. **4**(2): p. 17-29.
- 595 27. Dworkin, R.H., et al., *Development and initial validation of an expanded and revised* 596 *version of the Short-form McGill Pain Questionnaire (SF-MPQ-2).* Pain, 2009. **144**(1-2): 597 p. 35-42.
- 598 28. Beck, A.T., et al., *Beck-Depressions-Inventar Revision. Deutsche Adaption.* © 2006 599 Harcourt Test Services GmbH, Frankfurt/M. 2. Auflage © 2009 Pearson Assessment 600 & Information GmbH, Frankfurt am Main.



# Appendix 1: Schedule of assessments

| Time (days) | >-1<br>day | 0 | +7 | +14 | +28 | +35 | +42 | +56 | +63 | +70 | +84 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Informati<br>on | Infusion<br>1 | Questionn<br>aires<br>online | Questionn<br>aires<br>online | Infusion<br>2 | Questionn<br>aires<br>online | Questionn<br>aires<br>online | Infusion<br>3 | Questionn<br>aires<br>online | Questionn<br>aires<br>online | Questionn<br>aires<br>online |
| oral and written<br>Information | + | | | | | | | | | | |
| Written consent | + | | | | | | | | | | |
| check inclusion-/<br>exclusion criteria | + | | | | | | | | | | |
| Medical history | + | | | | | | | | | | |
| Participant<br>Characteristics | | + | | | | | | | | | |
| Questionnaires<br>Side effects | | + | | | + | | | + | | | |
| Blood Sampling | | + | | | + | | | + | | | |
| Short form McGill | | + | + | + | + | + | + | + | + | + | + |
| Beck Depression | | + | + | + | + | + | + | + | + | + | + |

